CLINICAL TRIAL: NCT07329595
Title: Monitoring the Clinical and Immunological Effects of Microbiome Changes Following Severe Burn Injury
Acronym: microbiome
Status: Recruiting | Type: Observational
Sponsor: Tamas Vegh, MD (Other)
Responsible Party: Sponsor-Investigator, Tamas Vegh, MD, MD PhD, University of Debrecen
Organization: University of Debrecen (Other)
Other Study IDs: AITT 2023/5; RKEB/IKEB 6649/2023 (Registry Identifier: Regional and Institutional Ethics Committee University of Debrecen Clinical Center); NNGYK/15506-5/2024 (Registry Identifier: National Centre for Public Health and Pharmacy)
Record Dates: First submitted 2025-11-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Severely Burned Patients; Gut Microbiota Diversity and Composition; Inflammatory Responses
Keywords: severe burn injury; gut microbiome
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to longitudinally monitor dynamic changes in the gut microbiome following severe burn injury using fecal samples. Under standard nutritional protocols and intensive care management, serial fecal sampling is performed to assess alterations in microbiome diversity and composition, as well as the indirect effects of these changes on measurable inflammatory biomarkers, endocrine, hematological, immunological, and other organ-specific parameters, the clinical course, and patient outcomes.

DETAILED DESCRIPTION:
Severe burn injury induces stress-related intestinal damage, leading to decreased gut perfusion, cellular injury, increased mucosal permeability, and reduced intestinal motility. These pathophysiological changes facilitate bacterial and endotoxin translocation, making the gut microbiome a major source of endogenous infection. Recent evidence indicates that the gut microbiome plays a critical role in regulating immune responses and supporting post-injury recovery, while also contributing to the development of complications such as sepsis and multi-organ failure.

The aim of this study is to longitudinally monitor dynamic changes in the gut microbiome following severe burn injury using fecal samples. Under standard nutritional protocols and intensive care management, serial fecal sampling is performed to assess alterations in microbiome diversity and composition, as well as the indirect effects of these changes on measurable inflammatory biomarkers, endocrine, hematological, immunological, and other organ-specific parameters, the clinical course, and patient outcomes. Clinical outcomes are evaluated based on mortality, length of hospital stay, duration of mechanical ventilation, incidence of secondary infections, rate of bacteremia, organ failure and its severity (assessed using the SOFA score), and wound healing.

Upon enrollment, patients undergo rectal swab collection and initial fecal sampling, followed by weekly fecal sample collection one to two times per week, alongside weekly laboratory investigations in addition to standard care. For microbiome analysis, DNA is extracted from fecal samples, followed by PCR amplification of the 16S bacterial rRNA operon. The amplified regions are sequenced, and taxa are identified based on sequence data. Relative abundances of taxa are calculated, and alpha- and beta-diversity metrics are compared within serial samples from individual patients and between patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age between 18 and 65 years) meeting the diagnostic criteria for severe burn injury, burns involving more than 20% of the total body surface area (TBSA) and/or inhalation injury.
* Burn injury caused by scalding, flame, electrical, contact, or chemical exposure
* Hospital admission within 24 hours following injury

Exclusion Criteria:

* Patients with inflammatory bowel diseases or malignant neoplasms.
* Patients with a history of major gastric and/or intestinal resections
* Patients in a pre-injury ECOG performance status of 4.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty adult patients (age between 18 and 65 year) meeting the diagnostic criteria for severe burn injury, burns involving more than 20% of the total body surface area (TBSA) and/or inhalation injury. Burn injury caused by scalding, flame, electrical, contact, or chemical exposure. Hospital admission within 24 hours following injury.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The abundance and bio-diversity of gut microbiota | Day of admission, one to two times per week up to 12 weeks
  Genomic DNA is extracted from the collected samples, followed by PCR amplification of the eubacterial 16S rRNA gene. The amplified region is subsequently sequenced, and taxonomic assignment is performed based on sequence analysis. Following the calculation of relative taxonomic abundances, alpha and beta diversity metrics are compared across longitudinal samples within individual patients and between patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lenke Jenei Kluch, MD, Principal Investigator — University of Debrecen
Locations (1):
- University of Debrecen, Department of Anesthesiology and Intensive Care, Debrecen, Hajdú-Bihar, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nakajima M, Kojiro M, Aso S, Matsui H, Fushimi K, Kaita Y, Goto H, Yamaguchi Y, Yasunaga H. Effect of high-dose vitamin C therapy on severe burn patients: a nationwide cohort study. Crit Care. 2019 Dec 12;23(1):407. doi: 10.1186/s13054-019-2693-1. PMID 31831039
- [Background] Song MJ, Kim S, Boo D, Park C, Yoo S, Yoon HI, Cho YJ. Comparison of proton pump inhibitors and histamine 2 receptor antagonists for stress ulcer prophylaxis in the intensive care unit. Sci Rep. 2021 Sep 16;11(1):18467. doi: 10.1038/s41598-021-98069-7. PMID 34531488
- [Background] Tanaka H, Matsuda T, Miyagantani Y, Yukioka T, Matsuda H, Shimazaki S. Reduction of resuscitation fluid volumes in severely burned patients using ascorbic acid administration: a randomized, prospective study. Arch Surg. 2000 Mar;135(3):326-31. doi: 10.1001/archsurg.135.3.326. PMID 10722036
- [Background] Wischmeyer PE. Nutrition Therapy in Sepsis. Crit Care Clin. 2018 Jan;34(1):107-125. doi: 10.1016/j.ccc.2017.08.008. Epub 2017 Oct 13. PMID 29149933
- [Background] Wald EL, Badke CM, Hintz LK, Spewak M, Sanchez-Pinto LN. Vitamin therapy in sepsis. Pediatr Res. 2022 Jan;91(2):328-336. doi: 10.1038/s41390-021-01673-6. Epub 2021 Jul 31. PMID 34333556
- [Background] Kahn SA, Beers RJ, Lentz CW. Resuscitation after severe burn injury using high-dose ascorbic acid: a retrospective review. J Burn Care Res. 2011 Jan-Feb;32(1):110-7. doi: 10.1097/BCR.0b013e318204b336. PMID 21131846
- [Background] Jeschke MG, Gauglitz GG, Kulp GA, Finnerty CC, Williams FN, Kraft R, Suman OE, Mlcak RP, Herndon DN. Long-term persistance of the pathophysiologic response to severe burn injury. PLoS One. 2011;6(7):e21245. doi: 10.1371/journal.pone.0021245. Epub 2011 Jul 18. PMID 21789167
- [Background] Wang Y, Shu Z, Zhu W, Zhou L, Song H, Luo G. The Prognostic Value of N-Terminal pro-Brain Natriuretic Peptide (NT-proBNP) in Major Burn Patients With Sepsis. J Burn Care Res. 2022 Nov 2;43(6):1351-1357. doi: 10.1093/jbcr/irac037. PMID 35303085
- [Background] Moreno R, Rhodes A, Piquilloud L, Hernandez G, Takala J, Gershengorn HB, Tavares M, Coopersmith CM, Myatra SN, Singer M, Rezende E, Prescott HC, Soares M, Timsit JF, de Lange DW, Jung C, De Waele JJ, Martin GS, Summers C, Azoulay E, Fujii T, McLean AS, Vincent JL. The Sequential Organ Failure Assessment (SOFA) Score: has the time come for an update? Crit Care. 2023 Jan 13;27(1):15. doi: 10.1186/s13054-022-04290-9. PMID 36639780
- [Background] McClave SA, Patel J, Bhutiani N. Should fecal microbial transplantation be used in the ICU? Curr Opin Crit Care. 2018 Apr;24(2):105-111. doi: 10.1097/MCC.0000000000000489. PMID 29432297
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Fu Y, Moscoso DI, Porter J, Krishnareddy S, Abrams JA, Seres D, Chong DH, Freedberg DE. Relationship Between Dietary Fiber Intake and Short-Chain Fatty Acid-Producing Bacteria During Critical Illness: A Prospective Cohort Study. JPEN J Parenter Enteral Nutr. 2020 Mar;44(3):463-471. doi: 10.1002/jpen.1682. Epub 2019 Aug 6. PMID 31385326
- [Background] Schroeder BO, Birchenough GMH, Stahlman M, Arike L, Johansson MEV, Hansson GC, Backhed F. Bifidobacteria or Fiber Protects against Diet-Induced Microbiota-Mediated Colonic Mucus Deterioration. Cell Host Microbe. 2018 Jan 10;23(1):27-40.e7. doi: 10.1016/j.chom.2017.11.004. Epub 2017 Dec 21. PMID 29276171
- [Background] He W, Wang Y, Wang P, Wang F. Intestinal barrier dysfunction in severe burn injury. Burns Trauma. 2019 Jul 26;7:24. doi: 10.1186/s41038-019-0162-3. eCollection 2019. PMID 31372365
- [Background] Earley ZM, Akhtar S, Green SJ, Naqib A, Khan O, Cannon AR, Hammer AM, Morris NL, Li X, Eberhardt JM, Gamelli RL, Kennedy RH, Choudhry MA. Burn Injury Alters the Intestinal Microbiome and Increases Gut Permeability and Bacterial Translocation. PLoS One. 2015 Jul 8;10(7):e0129996. doi: 10.1371/journal.pone.0129996. eCollection 2015. PMID 26154283
- [Background] Lima KM, Davis RR, Liu SY, Greenhalgh DG, Tran NK. Longitudinal profiling of the burn patient cutaneous and gastrointestinal microbiota: a pilot study. Sci Rep. 2021 May 21;11(1):10667. doi: 10.1038/s41598-021-89822-z. PMID 34021204
- [Background] Pan YY, Fan YF, Li JL, Cui SY, Huang N, Jin GY, Chen C, Zhang C. [Analysis of the dynamic changes in gut microbiota in patients with extremely severe burns by 16S ribosomal RNA high-throughput sequencing technology]. Zhonghua Shao Shang Za Zhi. 2020 Dec 20;36(12):1159-1166. doi: 10.3760/cma.j.cn501120-20200518-00271. Chinese. PMID 33379852
- [Background] Feng Y, Huang Y, Wang Y, Wang P, Song H, Wang F. Antibiotics induced intestinal tight junction barrier dysfunction is associated with microbiota dysbiosis, activated NLRP3 inflammasome and autophagy. PLoS One. 2019 Jun 18;14(6):e0218384. doi: 10.1371/journal.pone.0218384. eCollection 2019. PMID 31211803
- [Background] Rousseau AF, Losser MR, Ichai C, Berger MM. ESPEN endorsed recommendations: nutritional therapy in major burns. Clin Nutr. 2013 Aug;32(4):497-502. doi: 10.1016/j.clnu.2013.02.012. Epub 2013 Mar 14. PMID 23582468
- [Background] Clark A, Imran J, Madni T, Wolf SE. Nutrition and metabolism in burn patients. Burns Trauma. 2017 Apr 17;5:11. doi: 10.1186/s41038-017-0076-x. eCollection 2017. PMID 28428966
- [Background] Rice TC, Armocida SM, Kuethe JW, Midura EF, Jain A, Hildeman DA, Healy DP, Gulbins E, Caldwell CC. Burn injury influences the T cell homeostasis in a butyrate-acid sphingomyelinase dependent manner. Cell Immunol. 2017 Mar;313:25-31. doi: 10.1016/j.cellimm.2016.12.004. Epub 2016 Dec 26. PMID 28063598
- [Background] Feng Y, Huang Y, Wang Y, Wang P, Wang F. Severe burn injury alters intestinal microbiota composition and impairs intestinal barrier in mice. Burns Trauma. 2019 Jul 4;7:20. doi: 10.1186/s41038-019-0156-1. eCollection 2019. PMID 31312663
- [Background] Sun M, Wu W, Chen L, Yang W, Huang X, Ma C, Chen F, Xiao Y, Zhao Y, Ma C, Yao S, Carpio VH, Dann SM, Zhao Q, Liu Z, Cong Y. Microbiota-derived short-chain fatty acids promote Th1 cell IL-10 production to maintain intestinal homeostasis. Nat Commun. 2018 Sep 3;9(1):3555. doi: 10.1038/s41467-018-05901-2. PMID 30177845
- [Background] Macfarlane GT, Macfarlane S. Fermentation in the human large intestine: its physiologic consequences and the potential contribution of prebiotics. J Clin Gastroenterol. 2011 Nov;45 Suppl:S120-7. doi: 10.1097/MCG.0b013e31822fecfe. PMID 21992950
- [Background] Korkmaz HI, Flokstra G, Waasdorp M, Pijpe A, Papendorp SG, de Jong E, Rustemeyer T, Gibbs S, van Zuijlen PPM. The Complexity of the Post-Burn Immune Response: An Overview of the Associated Local and Systemic Complications. Cells. 2023 Jan 17;12(3):345. doi: 10.3390/cells12030345. PMID 36766687
- [Background] Luck ME, Herrnreiter CJ, Choudhry MA. Gut Microbial Changes and their Contribution to Post-Burn Pathology. Shock. 2021 Sep 1;56(3):329-344. doi: 10.1097/SHK.0000000000001736. PMID 33481548
- [Background] Rae L, Fidler P, Gibran N. The Physiologic Basis of Burn Shock and the Need for Aggressive Fluid Resuscitation. Crit Care Clin. 2016 Oct;32(4):491-505. doi: 10.1016/j.ccc.2016.06.001. Epub 2016 Aug 2. PMID 27600122
- [Background] Jeschke MG, van Baar ME, Choudhry MA, Chung KK, Gibran NS, Logsetty S. Burn injury. Nat Rev Dis Primers. 2020 Feb 13;6(1):11. doi: 10.1038/s41572-020-0145-5. PMID 32054846